CLINICAL TRIAL: NCT06163885
Title: The Effect of Flipped Classroom and Peer-Supported Education on Nursing Students' Stoma Care Skills and Academic Self-Efficacy:A Randomized Controlled Study
Brief Title: The Effect of Flipped Classroom and Peer-Supported Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, Dr, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19785
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Stoma Colostomy; Self Efficacy
Keywords: flipped classroom; stoma care; peer-supported learning; academic self-efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peer-supported training group (Experimental): Peer-supported training groups consist of 36 people. Participants in this group will receive a four-hour stoma care skill training from their peers. The group's knowledge and skills in stoma care were evaluated by two independent observers
  Interventions: Other: Stoma care education with peer-supported education model
- flipped classroom training group (Experimental): flipped classroom training groups consist of 35 people. Participants in this group will receive a four-hour stoma care skill training from their educator. The group's knowledge and skills in stoma care were evaluated by two independent observers
  Interventions: Other: Stoma care education with flipped classroom
- Control group (No Intervention): Control training groups consist of 35 people. Participants in this group will receive a four-hour stoma care skill training from their educator. The group's knowledge and skills in stoma care were evaluated by two independent observers

INTERVENTIONS:
Other: Stoma care education with flipped classroom — Flipped classroom model will use for stoma care education.These training models will explore which of them will be most useful for participants in the acquisition of stoma care skills and knowledge. It will also monitor whether there is any change in the level of academic self-efficacy of nursing students who follow these educational models.
  Arms: flipped classroom training group
Other: Stoma care education with peer-supported education model — Peer-supported education model will use for stoma care education.These training models will explore which of them will be most useful for participants in the acquisition of stoma care skills and knowledge. It will also monitor whether there is any change in the level of academic self-efficacy of nursing students who follow these educational models.
  Arms: peer-supported training group

SUMMARY:
In the randomized controlled study, the aim is to compare the effect of flipped classroom, peer-supported and traditional education on the knowledge and skills of nursing students in stoma care and on academic self-efficacy.

The sample consisted of 106 nursing students who studied at the Nursing Faculty. The data was collected using the Personal Information Form, the Stoma Care Skill Rubric, Stoma care information form, and the Academic Self-Efficacy Scale in Nursing Undergraduate Students The data will be analyzed using the number, percentage, average, standard deviation, minimum, maximum, median, skewness and kurtosis, Mann-Whitney U Test, Spearman Rho Correlation Test.

DETAILED DESCRIPTION:
In the randomized controlled study, the aim is to compare the effect of flipped classroom, peer-supported and traditional education on the knowledge and skills of nursing students in stoma care and on academic self-efficacy.

The sample consisted of 106 nursing students who studied at the Nursing Faculty. The data was collected using the Personal Information Form, the Stoma Care Skill Rubric, Stoma care information form, and the Academic Self-Efficacy Scale in Nursing Undergraduate Students The data will be analyzed using the number, percentage, average, standard deviation, minimum, maximum, median, skewness and kurtosis, Mann-Whitney U Test, Spearman Rho Correlation Test.

The hypotheses of the research; H1: Flipped classroom and peer-supported training groups, stoma care information scores are higher than in the control group.

H2: Flipped classroom and peer-supported training groups have higher stoma care skill scores than the control group.

H3: The academic self-efficacy score of flipped classroom and peer-supported training groups increases after the initiative.

H4: There is a difference stoma care skill score between flipped classroom and peer-supported training groups H5: There is a difference stoma care knowledge score between flipped classroom and peer-supported training groups

Flipped classroom, one of the learner-centered education models, consists of a combination of web-based education and traditional education. Web-based recordings can be synchronous and asynchronous. The learner accesses the instruction provided by the educator via the internet. After the basic learning gained in the internet environment, the educator obtains high-level cognitive learning through face-to-face discussion, analysis and synthesis in the classroom environment.

Peer -supported education; It is the educating and motivating of peers (peer learners) by peer educators (peer counselors) who have similar characteristics such as age, education level, profession and interests, through formal or informal educational activities. Peer- -supported education has many benefits for the learner, such as taking responsibility, gaining group/team work skills, supporting psychomotor skill development, and increasing academic success.

Academic self-efficacy (ASE) is the individual's self-confidence and belief that he or she can accomplish an academic task. Self-efficacy increases or decreases depending on the individual's previous experiences of success, the experiences of others, and the verbal support he receives from others. In addition, the individual's physical and emotional state and stress level affect his sense of self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* to be enrolled in the Surgical Diseases Nursing course (stoma care skills are included in this course)
* Not previously trained in stoma care
* Not working as a part-time/full-time nurse

Exclusion Criteria:

* Not willing to participate in the study
* Previously trained in stoma care
* Having previously cared for a stoma
* Working part-time/full-time as a nurse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Academic self-efficacy | total 12 weeks
  Academic self-efficacy scores of the experimental groups change after the intervention

SECONDARY OUTCOMES:
Stoma Care Skill Score | total 12 weeks
  There is a difference between the experimental groups and the control group in terms of Stoma Care Skill Score

OTHER OUTCOMES:
Stoma Care Knowledge Score | total 12 weeks
  There is a difference between the experimental groups and the control group in terms of Stoma Care Skill Knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Olga İncesu, Dr, Principal Investigator — Istanbul University-Cerrahpaşa Florence Nightingale Faculty of Nursing
Locations (1):
- Florence Nightingale Faculty of Nursing, Istanbul, Şişli, Turkey (Türkiye)